CLINICAL TRIAL: NCT01951573
Title: Delefilcon A Multifocal Plus Power Lens Design Evaluation
Brief Title: Evaluation of a New Daily Disposable Multifocal Contact Lens Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C-13-011
Record Dates: First submitted 2013-09-24; First posted 2013-09-26 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Presbyopia; Hyperopia; Refractive Error
Keywords: contact lenses; multifocal; daily disposable; silicone hydrogel; presbyopia
MeSH Terms: conditions — Presbyopia; Hyperopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delefilcon A MF, then AOAMF (Other): Delefilcon A multifocal contact lenses first, followed by lotrafilcon B multifocal contact lenses. Each product worn bilaterally (ie, in both eyes) for 9-12 hours, with a 1-8 day washout separating the 2 wear periods.
  Interventions: Device: Delefilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses
- AOAMF, then Delefilcon A MF (Other): Lotrafilcon B multifocal contact lenses first, followed by delefilcon A multifocal contact lenses. Each product worn bilaterally (ie, in both eyes) for 9-12 hours, with a 1-8 day washout separating the 2 wear periods.
  Interventions: Device: Delefilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses

INTERVENTIONS:
Device: Delefilcon A multifocal contact lenses — Silicone hydrogel multifocal contact lenses for daily wear, daily disposable use
Device: Lotrafilcon B multifocal contact lenses — Silicone hydrogel multifocal contact lenses with a labeled indication for daily wear and extended wear use of up to 6 days with monthly replacement
  Other Names: AIR OPTIX® AQUA MULTIFOCAL

SUMMARY:
The purpose of this study is to demonstrate non-inferiority of a new daily disposable multifocal contact lens in plus powers against the commercially available AIR OPTIX® AQUA MULTIFOCAL (AOAMF) lens in high contrast/high illumination (HC/HI) near visual acuity (VA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal eyes who are not using any ocular medication.
* Must sign the Informed Consent document.
* Habitual lens power within the range available for the study lenses (+1.00 to +3.50 diopters(D)).
* Manifest cylinder less than or equal to 0.75D.
* Best corrected distance VA greater than or equal to 20/25 in each eye.
* Existing soft contact lens (CL) wearers who wear contact lenses in both eyes at least 5 days per week.
* Presbyopic with a spectacle addition (ADD) >0.50D and <2.75D.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular disease, inflammation, or abnormality that contraindicates CL wear.
* Any use of systemic or ocular medications for which CL wear could be contraindicated.
* History of herpetic keratitis.
* History of refractive surgery or irregular cornea.
* A clinically significant dry eye that precludes CL wear.
* Participation of the subject in a clinical study (including CL or CL care product) within the previous 30 days.
* Monocular (only 1 eye with functional vision).
* History of intolerance or hypersensitivity to any component of the test articles.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Nick, Dipl. Ing., Study Director — CIBA VISION GmbH

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the US.
Pre-assignment Details: Of the 36 enrolled, 2 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (34).
Groups:
- Delefilcon A MF, Then AOAMF; AOAMF, Then Delefilcon A MF: Each product worn bilaterally (ie, in both eyes), as randomized, for 9-12 hours, with a 1-8 day washout separating the 2 wear periods.
Period: Period 1, First 9 Hours of Wear
Arm/Group | Delefilcon A MF, Then AOAMF | AOAMF, Then Delefilcon A MF
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Delefilcon A MF, Then AOAMF | AOAMF, Then Delefilcon A MF
Started | 17 | 17
Completed | 17 | 16
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2, Second 9 Hours of Wear
Arm/Group | Delefilcon A MF, Then AOAMF | AOAMF, Then Delefilcon A MF
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any Investigational Product (IP) evaluated in this study.
Groups:
- Overall: Delefilcon A MF and AOAMF contact lenses worn during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: High Contrast/High Illumination (HC/HI) Binocular Visual Acuity (VA) at Near
Description: Near VA was assessed binocularly (both eyes together) at 40 centimeters, with over-refraction (OR), if necessary, and measured in logMAR units (logarithm of the minimum angle of resolution). A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity, with a negative value denoting better than 20/20 visual acuity.
Time Frame: Dispense (Day 1), Hour 9
Population: This analysis population includes all randomized subjects excluding those who met any of the specified deviation criteria.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Delefilcon A MF; AOAMF: Contact lenses worn during Period 1 or Period 2 for 9-12 hours
Arm/Group | Delefilcon A MF | AOAMF
Number analyzed (Participants) | 33 | 34
logMAR
  Dispense | 0.10 (0.09) | 0.12 (0.06)
  Hour 9 | 0.08 (0.09) | 0.09 (0.07)

2. Secondary Outcome: HC/HI Binocular VA at Distance
Description: Distance VA was assessed binocularly (both eyes together) at 6 meters, with over-refraction (OR), if necessary, and measured in logMAR units (logarithm of the minimum angle of resolution). A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity, with a negative value denoting better than 20/20 visual acuity.
Time Frame: Dispense (Day 1), Hour 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Delefilcon A MF | AOAMF
Number analyzed (Participants) | 33 | 34
logMAR
  Dispense | -0.02 (0.06) | -0.03 (0.06)
  Hour 9 | 0.00 (0.07) | -0.01 (0.07)

3. Secondary Outcome: Over-refraction (OR) Monocular at Distance
Description: OR (the amount of additional correction needed to improve VA) at distance (equivalent to 6 meters) was assessed monocularly (for each eye separately) in diopters (D). Both eyes contributed to the mean.
Time Frame: Dispense (Day 1), Hour 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Diopters
Units Other Than Participants: eyes
Arm/Group | Delefilcon A MF | AOAMF
Number analyzed (Participants) | 33 | 34
Number analyzed (eyes) | 66 | 68
Diopters
  Dispense | 0.00 (0.00) | 0.00 (0.00)
  Hour 9 | 0.11 (0.16) | 0.09 (0.14)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from 04 Oct 2013 to 12 Nov 2013. This analysis group includes all subjects/eyes exposed to any Investigational Product (IP) evaluated in this study.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device.
Arm/Group | Delefilcon A MF | AOAMF
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/33 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes